CLINICAL TRIAL: NCT06888518
Title: Building Up the Vaginal Flora Using Multistrain Probiotics in Patients with Bacterial Vaginosis
Brief Title: Multistrain Probiotics Against Bacterial Vaginosis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Institut AllergoSan Pharma GmbH (Industry)
Collaborators: Medical University of Vienna (Other); MEDIZINISCHE UNIVERSITAT GRAZ (Unknown); Medizinische Universität Innsbruck, OE Clinical Trial Center (Koordinierungszentrum für klinische Studien, KKS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Gruber_BV_Floraplus; Institute AllergoSan (Other: Institute AllergoSan)
Record Dates: First submitted 2025-02-25; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Bacterial Vaginosis (BV)
Keywords: Bacterial vaginosis; vaginal dysbiosis; probiotics
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Probiotics; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, multicenter study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotic dietary supplement (Active Comparator): twice daily probiotic OMNi-BiOTiC® FLORA plus+ plus antibiotic treatment
  Interventions: Dietary Supplement: OMNi-BiOTiC® FLORA plus+; Drug: antibiotic
- controll group (Other): antibiotic treatment without probiotics
  Interventions: Drug: antibiotic

INTERVENTIONS:
Dietary Supplement: OMNi-BiOTiC® FLORA plus+ — specially selected probiotic strains for the diatary treatment of Lactobacillus deficiencies in women
  Other Names: probiotic
  Arms: probiotic dietary supplement
Drug: antibiotic — regular antibiotic treatment against bacterial vaginosis
  Other Names: antibiotic treatment

SUMMARY:
The primary aim of the study is to clarify whether and to what extent the consumption of the multistrain probiotic OMNi-BiOTiC® FLORA plus+ has a positive effect on the vaginal flora and reduces BV. This is determined using the Nugent score and the blackbird criteria.

In one subgroup, the composition of the vaginal microbiome is analysed using 16S rRNA gene sequencing.

DETAILED DESCRIPTION:
If bacterial vaginosis (BV) is detected using the Nugent score (= gold standard for studies) and Amsel criteria, the patient in question is eligible for the study, provided the following additional criteria are met:

* >16 years of age
* Proof of BV using the Nugent Score (≥ 6)
* Written informed consent for the study (the document is available in printed form in the study folder). Additional parental information is available for underage patients

Please also note the following exclusion criteria:

* Consumption of other probiotics within the last 4 weeks
* Pregnancy, breastfeeding
* Infections of the urogenital tract
* Participation in another study
* Infection with other vaginal germs or vaginal mycosis
* Hepatitis B, C or HIV infection
* Planned hospitalisation during the intervention period After clarification of the inclusion and exclusion criteria and consent to participate in the study on the part of the patient (signed declaration of consent), the patient is included in the study. The patient is prescribed an antibiotic (oral or topical) according to the guidelines for the treatment of BV. Based on a randomisation list with consecutive numbers provided by us, the patient is allocated to the OMNi-BiOTiC® FLORA plus+ group (they take the AB + probiotic) or to the control group (only receive the antibiotic). This ensures proper, random allocation to the respective group.

The doctor fills in part 1 of the questionnaire on BV symptoms together with the patient. The patients in the probiotics group are given OMNi-BiOTiC® FLORA plus+ by the doctor (2 packs per patient; provided by the AllergoSan Institute), which is to be taken twice a day for 4 weeks. The control group is only prescribed the antibiotic (we do not prescribe an AB - the doctor decides which AB).

After four weeks of the study, the patients return to the gynaecologist's practice for a follow-up visit. The Nugent Score and Amsel criteria are determined again and part 2 of the questionnaire is completed together with the doctor. The study is then completed for the patient.

Optional: Some of the patients will also have a vaginal swab taken for microbiome analysis (30 patients; 15 from the AB+ probiotics group, 15 from the control group). This swab is taken by the doctor at study inclusion and after 4 weeks of the study. The samples (vaginal swabs) are stored in the refrigerator until they are collected.

ELIGIBILITY:
Inclusion Criteria:

* 16 years
* Proof of BV using the Nugent Score (> 6)
* Written informed consent for the study (the document is available in printed form in the study folder).
* Additional parental information is available for underage patients

Exclusion Criteria:

* Consumption of other probiotics within the last 4 weeks
* Pregnancy, breastfeeding
* Infections of the urogenital tract
* Participation in another study
* Infection with other vaginal germs or vaginal mycosis
* Hepatitis B, C or HIV infection
* Planned hospitalisation during the intervention period

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
reduction of patients with BV | 4 weeks
  the primary endpoint is the reduction in the number of patients with BV (defined as Nugent Score >6) in the probiotic group compared to the control group

SECONDARY OUTCOMES:
vaginal swab and general well-being | 4 weeks
  The Nugent Score and the Amsel criteria before (vaginal pH>4.5, presence of >20% per HPF of "clue cells" on wet mount examination, positive amine or "whiff" test, homogeneous, non-viscous, milky-white discharge adherent to the vaginal walls) and after treatment (vaginal swab), the general well-being of the test subjects (questionnaire), the improvement in the symptoms of BV (itching, burning, etc.), the number of days of treatment with antibiotics and, in a subgroup, the differences in the composition of the vaginal microbiome using 16S rRNA sequencing (alpha- and betadiversity) are recorded as secondary target variables.
  In addition, compliance and tolerability of the preparation, including side effects, are examined.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Maria Gruber, Univ. Prof. Dr., Principal Investigator — Wahlarztordination Wien, Lainzerstrasse 147, A-1130 Wien
Locations (1):
- Wahlarzpraxis, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Because study was terminated prematurely